CLINICAL TRIAL: NCT00928915
Title: Multicenter, Prospective Randomized Trial on the Use of Prothrombin Complex and Fresh Frozen Plasma in Patients With Intracerebral Hemorrhage Related to Vitamin K Antagonists
Brief Title: International Normalized Ratio (INR) Normalization in Coumadin Associated Intracerebral Haemorrhage
Acronym: INCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Thorsten Steiner, Prof. Dr., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFmu-344/2008; EUDRAT 2008-005653-37
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Intracranial Hemorrhages
Keywords: Intracranial Hemorrhages; Vitamin-K antagonist; Hemostatic treatment; Prothrombin complex; Fresh frozen plasma; Intracranial Hemorrhages related to vitamin-K antagonist
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prothrombin complex concentrate (PCC) (Experimental): intravenously, 30 IU/kg
  Interventions: Drug: Prothrombin complex concentrate (PCC); fresh frozen plasma (FFP)
- Fresh frozen plasma (FFP) (Experimental): intravenously, 20ml/kg
  Interventions: Drug: Prothrombin complex concentrate (PCC); fresh frozen plasma (FFP)

INTERVENTIONS:
Drug: Prothrombin complex concentrate (PCC); fresh frozen plasma (FFP) — intravenous, repeated until INR ≤ 1.2

SUMMARY:
Intracerebral haemorrhage (ICH) is the most feared complication in patients on vitamin K antagonists (VKA). VKA related ICH occurs 8-10 times more frequently and the mortality is 2 times higher than in non-anticoagulated patients. Mortality may rise up to 67%. The higher mortality rate may in part be due to the higher rate of haematoma expansion (HE) over a longer period after symptom onset. International guidelines recommend treatment of VKA-ICH with prothrombin complex (PCC) or fresh-frozen plasma (FFP) both in combination with Vitamin-K. But these recommendations are not based on randomized controlled trials. It is known that these drugs lower the INR, and thus it is assumed that normalization of coagulopathy may lead to haemostasis and reduction of HE. Safety and efficacy of these treatments have never been studied in a prospective controlled trial.

The investigators' questions are: How potent are PCC and FFP in normalization of the INR? What is the safety profile of each of these drugs?

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous ICH (intraparenchymal), subdural hematoma (SDH) diagnosed by CT scanning ≤ 12 hours after onset of symptoms. In case of unknown time of symptom onset: time between last seen in healthy condition and first CCT ≤ 12 hours.
* Therapy receiving vitamin K antagonists (VKA)
* International Normalized Ratio (INR) ≥ 2
* Signed informed consent form, or signed informed consent by a legal representative, judicial consent in cases where no legal representative is available in time, or consent of an independent physician familiar with the indication in cases where the first three possibilities can not be realized.

Exclusion Criteria:

* Patients with ICH not related to vitamin-K antagonist therapy or
* Patients with secondary ICH related to infarction, hemophilia or other coagulopathy, tumor, hemorrhagic infarction, cerebrovenous thrombosis, aneurysm, arteriovenous malformations (AVM) or severe trauma
* Deep Coma (GCS ≤ 5) at the time of admission or before intubation if intubated outside the hospital
* Known previous disability (mRS > 2 before stroke occurred)
* Acute myocardial ischemia, acute septicemia, acute crush injury, any history of acute hemorrhagic disseminated intravascular coagulation, acute thrombotic stroke
* Known history of intermittent claudication
* Known recent thrombotic event < 30 days
* Acute or known congestive heart failure (NYHA III, IV)
* Pulmonary edema
* Known liver failure (child-pugh-score C)
* Known alcohol or other drug abuse
* Known active malignant disease
* Known thrombocytopenia (platelets <50,000/µL), hemorrhagic diathesis (primary defects of coagulation, fibrinolysis, platelets)
* History of hypersensitivity to the investigational products or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational product
* Known allergy to heparin or history of heparin induced thrombocytopenia.
* Pregnancy and lactation
* Concomitant use of antithrombotic (with PTT > 1.5 of normal PTT), thrombolytic treatment.
* Use of aspirin, clopidogrel or dipyridamole or combinations thereof (e.g. Aggrenox®) is not an exclusion criterion. These drugs should be discontinued and not restarted earlier than 24 hours after normalization of INR if indicated.
* Previous participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
INR ≤ 1.2 within 3 hours after start of drug infusion | 3 hours

SECONDARY OUTCOMES:
Safety: Number of thromboembolic events | 90 days
Efficacy: Percentage of volume increase | 24 hours
Clinical outcome | day 90

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Steiner, MR, PhD, MME, Principal Investigator — Department of Neurology, Heidelberg University Hospital Germany
Locations (1):
- Heidelberg University Clinic, Heidelberg, Germany

REFERENCES:
- [Background] Steiner T, Griebe M, Ivandic B, et al. Multicenter, prospective randomized trial on the use of prothrombin complex and fresh frozen plasma to normalize the INR in patients with coumadine related intracerebral hemorrhage related to vitamin K antagonists - The INCH-trial. Cerebovascular Disease 2009;27:185
- [Background] Steiner T, Freiberger A, Griebe M, Husing J, Ivandic B, Kollmar R, Pfefferkorn T, Wartenberg KE, Weimar C, Hennerici M, Poli S. International normalised ratio normalisation in patients with coumarin-related intracranial haemorrhages--the INCH trial: a randomised controlled multicentre trial to compare safety and preliminary efficacy of fresh frozen plasma and prothrombin complex--study design and protocol. Int J Stroke. 2011 Jun;6(3):271-7. doi: 10.1111/j.1747-4949.2010.00560.x. Epub 2011 Jan 10. PMID 21557816
- [Result] Steiner T, Poli S, Griebe M, Husing J, Hajda J, Freiberger A, Bendszus M, Bosel J, Christensen H, Dohmen C, Hennerici M, Kollmer J, Stetefeld H, Wartenberg KE, Weimar C, Hacke W, Veltkamp R. Fresh frozen plasma versus prothrombin complex concentrate in patients with intracranial haemorrhage related to vitamin K antagonists (INCH): a randomised trial. Lancet Neurol. 2016 May;15(6):566-73. doi: 10.1016/S1474-4422(16)00110-1. Epub 2016 Apr 11. PMID 27302126
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112